CLINICAL TRIAL: NCT04433585
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3471851 (NKTR-358) in Adults With Systemic Lupus Erythematosus
Brief Title: A Study of LY3471851 in Adults With Systemic Lupus Erythematosus (SLE)
Acronym: ISLAND-SLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17422; J1P-MC-KFAJ (Other: Eli Lilly and Company); 2019-003323-38 (EudraCT Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: T regulatory cells (Tregs); Interleukin 2; Interleukin-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3471851 High Dose (Experimental): LY3471851 administered subcutaneously (SC).
  Interventions: Drug: LY3471851
- LY3471851 Mid Dose (Experimental): LY3471851 administered SC.
  Interventions: Drug: LY3471851
- LY3471851 Low Dose (Experimental): LY3471851 administered SC
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — Administered SC
  Other Names: Rezpegaldesleukin; REZPEG; NKTR-358
  Arms: LY3471851 High Dose; LY3471851 Low Dose; LY3471851 Mid Dose
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug LY3471851 (NKTR-358) is safe and effective in adults with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
LY3471851 is a potential first-in-class therapeutic that may address an underlying immune system imbalance in people with many autoimmune conditions. It targets the interleukin (IL-2) receptor complex in the body in order to stimulate proliferation of inhibitory immune cells known as regulatory T cells. By activating these cells, LY3471851 may act to bring the immune system back into balance.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of SLE at least 24 weeks prior to screening.
* Have documentation of having met at least 4 of 11 Revised Criteria for Classification of Systemic Lupus Erythematosus according to the 1997 Update of the 1982 American College of Rheumatology (ACR) criteria for classification of SLE prior to randomization.
* Have a positive antinuclear antibody (ANA) (titer ≥1:80) and/or a positive anti-double-stranded deoxyribonucleic acid (dsDNA), and/or a positive anti-Smith (anti-Sm) as assessed by a central laboratory during screening.
* Have a total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥6 during screening.
* Have a clinical SLEDAI-2K score ≥4 at randomization.
* Have active arthritis and/or active rash.

Exclusion Criteria:

* Have severe active lupus nephritis.
* Have active central nervous system (CNS) lupus.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (112):
- United States (23):
  - University of California - San Diego, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Stanford University Hospital, Stanford, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Great Neck, New York
  - NYU Langone, New York, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Accurate Clinical Management, Baytown, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Accurate Clinical Research, Houston, Texas
  - Fort Bend Clinical Research, LLC, Sugar Land, Texas
  - University of Washington Medical Center, Seattle, Washington
- Argentina (8):
  - DOM- Centro de Reumatologia, CABA, Buenos Aires
  - Centro Privado de Medicina Familiar / Mindout Research, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - APRILLUS Asistencia E Investigacion de Arcis Salud, CABA, Ciudad Autónoma de Buenos Aire
  - Clinica Adventista Belgrano, CABA, Ciudad Autónoma de Buenos Aire
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Hospital J. M. Ramos Mejía, Ciudad Autónoma de Buenos Aire
  - Hospital Córdoba, Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER-San Juan, San Juan
- Emeritus Research, Camberwell, Victoria, Australia
- University of Calgary, Calgary, Alberta, Canada
- Czechia (2):
  - INREA s.r.o., Ostrava, Ostrava Město
  - Revmatologicky ustav, Prague, Praha, Hlavní Mešto
- Germany (6):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universtitätsklinikum Essen AöR, Essen, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet, Herne, North Rhine-Westphalia
  - Klinikum Bad Bramstedt GmbH, Bad Bramstedt, Schleswig-Holstein
  - Universitätsklinikum Köln, Cologne
  - Klinik für Innere Medizin I, Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Hungary (3):
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Gyula, Bekes County
  - Qualiclinic, Budapest
  - Debreceni Egyetem Orvos-es Egészsegtudomanyi Centrum, Debrecen
- India (13):
  - Krishna Institute of Medical Science, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatanam, Andhra Pradesh
  - Amber Clinic, Ahmedabad, Gujarat
  - Swastik Rheumatology Clinic, Ahmedabad, Gujarat
  - Sushruta Multispeciality Hospital & Research Centre, Hubli, Karnataka
  - Government Medical College (GMC) Aurangabad, Aurangabad, Maharashtra
  - Government Medical College, Nagpur, Maharashtra
  - Jasleen Hospital, Nagpur, Maharashtra
  - All India Institute of Medical Sciences - Nagpur, Nagpur, Maharashtra
  - Sancheti Institute for Orthopaedics & Rehabilitation, Pune, Maharashtra
  - Center for Rheumatic Diseases, Pune, Maharashtra
  - Sancheti HealthCare Academy, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
- Israel (4):
  - Sheba Medical Center, Ramat Gan, Central District
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (12):
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - National Hospital Organization Chibahigashi National Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Okayama University Hospital, Okayama
  - Daini Osaka Police Hospital, Osaka
  - St. Luke's International Hospital, Tokyo
  - Keio university hospital, Tokyo
- Mexico (6):
  - CIMAB SA de CV, Torreón, Coahuila
  - Centro Medico del Angel, Mexicali, Estado de Baja California
  - Centro Integral en Reumatologia, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - RM Pharma Specialists S.A. de C.V., Mexico City, Mexico City
  - Clinica para el Diagnostico y Tratamiento de la Enfermedades, Mexico City, Mexico City
- Poland (4):
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Nova Reuma Społka Partnerska, Bialystok, Podlaskie Voivodeship
  - Nzoz Bif-Med, Bytom, Silesian Voivodeship
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
- Puerto Rico (4):
  - Centro Reumatologico Caguas, Caguas, PR
  - Latin Clinical Trial Center, San Juan, PR
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Mindful Medical Research, San Juan, PR
- Romania (4):
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - SC Centrul Medical Sana SRL, Bucharest
  - Spitalul Clinic Sf Maria Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei, Galati
- Russia (4):
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk, Kareliya, Respublika
  - Moscow City Clinical Hospital Number 15, Moscow, Moscow
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - Ryazan Regional Clinical Cardiology Dispensary, Ryazan
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Korea
  - Kyung Hee University Hospital, Seoul, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul, Seoul, Korea
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Quiron Infanta Luisa, Seville
- Taiwan (4):
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Ukraine (6):
  - Regional Clinical Hospital Center for Emergency medical care, Kharkiv
  - Edelweiss Medics LLC, Kyiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Multifield Medical Center of Odesa NMU (University Clinic#1), Odesa
  - Vinnytsya Regional Clinical Hospital, Vinnytsia
  - Regional Clinical Hospital of Zaporizhzhia, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3471851 in Adults With Systemic Lupus Erythematosus (SLE) (ISLAND-SLE) — https://trials.lillytrialguide.com/en-US/trial/2NrKmN7Zwj52k3UG9QrLqS

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a 24-week treatment period: participants randomly received either high dose LY3471851 or mid dose LY3471851 or low dose LY3471851 or placebo.
Groups:
- LY3471851 High Dose: Participants received a subcutaneous injection of high dose LY3471851 every 2 weeks from weeks 0 to 24.
- LY3471851 Mid Dose: Participants received a subcutaneous injection of mid dose LY3471851 every 2 weeks from weeks 0 to 24.
- LY3471851 Low Dose: Participants received a subcutaneous injection of low dose LY3471851 every 2 weeks from weeks 0 to 24.
- Placebo: Participants received a subcutaneous injection of placebo dose every 2 weeks from weeks 0 to 24.
Period: Overall Study
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
Started | 73 | 70 | 74 | 74
Completed | 44 | 57 | 55 | 65
Not Completed | 29 | 13 | 19 | 9
Not completed — Withdrawal by Subject | 15 | 3 | 15 | 6
Not completed — Adverse Event | 10 | 4 | 1 | 0
Not completed — Due to the conflict in Ukraine | 2 | 1 | 1 | 2
Not completed — Physician Decision | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo | Total
Number analyzed (Participants) | 73 | 70 | 74 | 74 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 69 | 74 | 72 | 287
  >=65 years | 1 | 1 | 0 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.4) | 41.3 (13.0) | 39.9 (12.0) | 41.6 (12.0) | 40.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 69 | 67 | 268
  Male | 5 | 6 | 5 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is based on responses from US sites only.
  Participants
    Hispanic or Latino | 9 | 11 | 4 | 11 | 35
    Not Hispanic or Latino | 5 | 3 | 11 | 5 | 24
    Unknown or Not Reported | 59 | 56 | 59 | 58 | 232
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 4 | 7 | 23
  Asian | 15 | 14 | 20 | 16 | 65
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 4 | 6 | 5 | 18
  White | 49 | 45 | 44 | 46 | 184
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 13 | 11 | 12 | 8 | 44
  Romania | 2 | 2 | 4 | 6 | 14
  Hungary | 0 | 1 | 0 | 1 | 2
  United States | 14 | 14 | 15 | 16 | 59
  Czechia | 1 | 0 | 1 | 3 | 5
  Japan | 6 | 3 | 6 | 4 | 19
  Ukraine | 10 | 7 | 8 | 10 | 35
  India | 8 | 8 | 12 | 10 | 38
  Spain | 1 | 1 | 0 | 0 | 2
  Russia | 1 | 3 | 0 | 1 | 5
  Canada | 1 | 0 | 0 | 0 | 1
  South Korea | 0 | 1 | 1 | 1 | 3
  Taiwan | 1 | 2 | 1 | 1 | 5
  Poland | 4 | 7 | 5 | 0 | 16
  Mexico | 7 | 9 | 8 | 12 | 36
  Israel | 1 | 0 | 0 | 1 | 2
  Australia | 0 | 0 | 1 | 0 | 1
  Germany | 3 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a ≥4 Point Reduction in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) 2000 (2K) Score at Week 24
Description: Percentage of Participants who Achieved a ≥4 Point Reduction in SLEDAI-2K Score at Week 24. A SLEDAI-4 response is defined as a ≥4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score from baseline. The SLEDAI-2K score range is from a minimum of 0 to a maximum of 105 (higher scores represent higher disease activity).
Time Frame: Week 24
Population: Modified Intent to Treat (mITT) patient population: All randomized patients with at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received a subcutaneous injection of placebo every 2 weeks from weeks 0 to 24.
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
Number analyzed (Participants) | 73 | 70 | 74 | 74
Participants | 20 | 27 | 22 | 22
Statistical Analysis 1: Comparison: LY3471851 Mid Dose vs Placebo; Test type: Superiority; p = 0.309, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.70 to 3.04]
Statistical Analysis 2: Comparison: LY3471851 Low Dose vs Placebo; Test type: Superiority; p = 0.944, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.47 to 2.03]
Statistical Analysis 3: Comparison: LY3471851 High Dose vs Placebo; Test type: Superiority; p = 0.649, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.40 to 1.78]

2. Secondary Outcome: Percentage of Participants Who Achieved British Isles Lupus Assessment Group (BILAG) Based Composite Lupus Assessment (BICLA) Response at Week 24.
Description: Percentage of Participants who Achieve BICLA Response at Week 24. The BILAG-based Composite Lupus Assessment (BICLA) is a composite index used to assess disease activity in SLE. A BICLA response is defined as:
  * Reduction of all baseline BILAG-2004 A to B or C or D; and baseline BILAG-2004 B to C or D; and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B.
  * No worsening from baseline in SLEDAI-2K, where worsening is defined as any increase from baseline in SLEDAI-2K.
  * No worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.30 points on a 3-point PGA visual analogue scale (VAS).
Time Frame: Week 24
Population: A subset of modified intent-to-treat (mITT) patients with at least 1 BILAG A score or 2 BILAG B scores at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
Number analyzed (Participants) | 60 | 56 | 59 | 60
Participants | 12 | 26 | 18 | 18
Statistical Analysis 1: Comparison: LY3471851 Mid Dose vs Placebo; Test type: Superiority; p = 0.131, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.83 to 4.30]
Statistical Analysis 2: Comparison: LY3471851 Low Dose vs Placebo; Test type: Superiority; p = 0.844, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.47 to 2.50]
Statistical Analysis 3: Comparison: LY3471851 High Dose vs Placebo; Test type: Superiority; p = 0.218, Regression, Logistic; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.24 to 1.39]

3. Secondary Outcome: Percentage of Participants Who Achieved Systemic Lupus Erythematosus Responder Index 4 (SRI-4) Response at Week 24
Description: Percentage of Participants who Achieved a SRI-4 Response at Week 24. A SRI-4 response is defined as a decrease in SLEDAI-2K >= 4 from baseline. No new BILAG A and no more than 1 new BILAG B disease activity score / organ domain (both compared with baseline), and no worsening in PGA (defined as an increase of 0.3 points [10 mm] from baseline.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
Number analyzed (Participants) | 73 | 70 | 74 | 74
Participants | 20 | 27 | 22 | 22
Statistical Analysis 1: Comparison: LY3471851 Low Dose vs Placebo; Test type: Superiority; p = 0.944, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.47 to 2.03]
Statistical Analysis 2: Comparison: LY3471851 Mid Dose vs Placebo; Test type: Superiority; p = 0.309, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.70 to 3.04]
Statistical Analysis 3: Comparison: LY3471851 High Dose vs Placebo; Test type: Superiority; p = 0.649, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.40 to 1.78]

4. Secondary Outcome: Percentage of Participants Who Achieved Lupus Low Disease Activity State (LLDAS) at Week 24
Description: Percentage of Participants who Achieved LLDAS at Week 24. A LLDAS response is defined as a low level of disease activity attained without use of low-dose steroids and/or standard-of-care immunosuppressant medications.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
Number analyzed (Participants) | 73 | 70 | 74 | 74
Participants | 12 | 18 | 11 | 10
Statistical Analysis 1: Comparison: LY3471851 Mid Dose vs Placebo; Test type: Superiority; p = 0.203, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.71 to 5.20]
Statistical Analysis 2: Comparison: LY3471851 Low Dose vs Placebo; Test type: Superiority; p = 0.865, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.38 to 3.16]
Statistical Analysis 3: Comparison: LY3471851 High Dose vs Placebo; Test type: Superiority; p = 0.896, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.38 to 3.05]

5. Secondary Outcome: Pharmacokinetics (PK): Trough Concentrations (Ctrough) of LY3471851
Description: LY3471851 plasma trough concentrations are the concentrations of drug in plasma immediately before the next dose is administered.
Time Frame: Week 24
Population: PK population at Week 24 is a subset of the mITT population with PK samples collected and available at Week 24.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose
Number analyzed (Participants) | 39 | 53 | 51
ng/mL | 214.4 (96.7) | 133.3 (50.6) | 55.9 (30.6)

ADVERSE EVENTS:
Time Frame: Adverse events will be reported from the time of the participant signing of the consent until 56 days after the last dose of study drug, up to a maximum of approximately 245 days (8 months). If randomized participants tested positive for antibody to hepatitis B core antigen (anti-HBc) at the screening visit, then the adverse events collection time frame is until 112 days after the last dose of study drug, up to a maximum of approximately 300 days (10 months).
Groups:
- LY3471851 Mid Dose; LY3471851 Low Dose: LY3471851 administered subcutaneously (SC).
- Placebo: Placebo administered subcutaneously (SC).
Arm/Group | LY3471851 High Dose | LY3471851 Mid Dose | LY3471851 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 1/70 | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 3/73 | 7/70 | 1/74 | 5/74
Other Adverse Events (participants affected / at risk) | 54/73 | 48/70 | 42/74 | 40/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LY3471851 High Dose (N=73) | LY3471851 Mid Dose (N=70) | LY3471851 Low Dose (N=74) | Placebo (N=74)
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LY3471851 High Dose (N=73) | LY3471851 Mid Dose (N=70) | LY3471851 Low Dose (N=74) | Placebo (N=74)
COVID-19 (Infections and infestations) | 3 | 8 | 4 | 5
Urinary tract infection (Infections and infestations) | 4 | 2 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 5 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 3 | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 2 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 11 | 7 | 3 | 0
Injection site reaction (General disorders) | 12 | 5 | 2 | 0
Fatigue (General disorders) | 6 | 1 | 3 | 0
Pain (General disorders) | 2 | 4 | 1 | 1
Injection site pruritus (General disorders) | 3 | 2 | 2 | 0
Asthenia (General disorders) | 3 | 1 | 0 | 1
Injection site erythema (General disorders) | 4 | 1 | 0 | 0
Injection site pain (General disorders) | 4 | 1 | 0 | 0
Injection site rash (General disorders) | 2 | 3 | 0 | 0
Injection site swelling (General disorders) | 2 | 1 | 0 | 0
Application site erythema (General disorders) | 0 | 2 | 0 | 0
Application site pruritus (General disorders) | 0 | 2 | 0 | 0
Application site reaction (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Administration site pain (General disorders) | 0 | 1 | 0 | 0
Application site inflammation (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 1 | 0 | 0
Injection site erosion (General disorders) | 1 | 0 | 0 | 0
Injection site exfoliation (General disorders) | 1 | 0 | 0 | 0
Injection site hypersensitivity (General disorders) | 1 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Mucosal ulceration (General disorders) | 0 | 1 | 0 | 0
Sensation of foreign body (General disorders) | 1 | 0 | 0 | 0
Swelling face (General disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Heart rate increased (Investigations) | 1 | 0 | 1 | 2
Urine protein/creatinine ratio increased (Investigations) | 1 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 1 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Urinary sediment (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 4 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 2
Cluster headache (Nervous system disorders) | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Ophthalmic migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 | 1 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04433585/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT04433585/SAP_001.pdf